CLINICAL TRIAL: NCT02984189
Title: Effect of Inspiratory Muscle Training Using the Critical Pressure on Recreational Cyclists: A Randomized Controlled Trial
Brief Title: Effect of Inspiratory Muscle Training on Recreational Cyclists
Acronym: IMT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Aparecida Maria Catai, Professor Aparecida Maria Catai, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 55990116.0.0000.5504
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Physical Exercise; Physical Therapy; Physical Performance; Critical Power; Respiratory Muscle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inspiratory Critical Pressure Group (Experimental): Inspiratory Critical Pressure will be used for training and will be determined, from a progressive inspiratory threshold-loading test will start with 50%MIP followed by 10%MIP increments, every 3min until subjects reached a load that there were unable to sustain for at least 1min (PThMAX). On another day, the subjects will perform a constant inspiratory loading test against a resistance of 95%, 100% and 105%PThMAX, for as long as they could tolerate. The intensity loads will be applied according the results of block randomization. The time elapsed until task failure was defined as inspiratory muscle endurance time, and will use to set the PThC. The respiratory work done (inspiratory pressure values) will be plotted in abscissa and the time-to-exhaustion in ordinate, and a linear regression going through the 3 points will be applied using the pressure-1/t relationship. The slope of the parallel line displaced downward projecting to the origin produce the PThC value.
  Interventions: Other: Inspiratory muscle training
- 60% Maximal Inspiratory Pressure Group (Active Comparator): 60% of maximal inspiratory pressure will be used for training.
  Interventions: Other: Inspiratory muscle training
- Sham Group (Sham Comparator): 6 cmH20 will be used for training.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — The inspiratory muscle training (IMT) will be realized, to compare three intensities differents the training (Inspiratory critical pressure, 60% maximal inspiratory pressure and sham). The IMT will be performed for 11 weeks (33 sessions, 3 times/week, 1-hour duration). The session will consist of 5-min warm-up (50% of the training load) and 3 sets of 15 minutes (breathing against 100% of the training load) with 1-min interval between them, using a linear inspiratory load resistor (Device: PowerBreathe K5).

SUMMARY:
Introduction: The inspiratory muscle training (IMT) has showed great benefits to the respiratory, autonomic system, and mainly to the improvement of physical performance in healthy subjects. The latter is related to the improvement of respiratory muscle strength, decreased of dyspnoea, peripheral fatigue and delay in activation of muscle metaboreflex during exercise. However, there is no consensus about the best training load to IMT, because the prescription has been done only using percentage of the maximal inspiratory pressure (MIP), and 60% of MIP has been the most used. Therefore, the IMT prescription protocol that takes into account the respiratory muscle strength and endurance can provide additional benefits to protocols commonly applied, once that respiratory muscle differs from the other muscles due to its greater muscle endurance. In the sense, the IMT using inspiratory critical pressure (PThC) comes up with an alternative, since the PThC calculation considers these characteristics. Objective:To evaluate the effect of the IMT, using PThC, on cardiovascular, respiratory, metabolic and autonomic responses in recreational cyclists and compare it to a IMT using 60% of MIP. Methods: Thirty men recreational cyclists (20-40 years), will be randomized to placebo group (PG, n = 10), PThC group (PTHCG, n = 10) and 60% of MIP group (60G, n = 10), taking into account the age and functional aerobic capacity. All subjects will perform the following evaluations: cardiovascular autonomic tests [heart rate variability (HRV) and blood pressure variability (BPV) at rest and after active postural change], pulmonary function testing, respiratory muscle strength (RMS) test, cardiopulmonary exercise testing (CPET), incremental respiratory muscle endurance test (iRME) [maximum respiratory pressure sustained for 1 minute (PThMAX)] and constant respiratory loads test (95%, 100% and 105% of PThMAX), both using an linear inspiratory load resistor (PowerBreathe K5). The PThC will be obtained from the linear regression using the time(TLIM) of and load of each constant test (95%, 100% and 105% PThMAX). During evaluations, the ECG (BioAmp FE132), blood pressure (BP), using Finometer Pro (Finapress Medical Systems) and respiration (Marazza) signals will be acquired. The signals will be coupled by data acquisition and analysis device (Power Lab 8/35) and sampled at 1000 Hz. Moreover, the oxyhemoglobin, deoxyhemoglobin and total hemoglobin responses will be measured by near-infrared spectroscopy (NIRS) (Oxymon MKIII), sampled at 250Hz. The IMT will be performed for 11 weeks (3 times/week, 1-hour duration). The session will consist of 5-min warm-up (50% of the training load) and 3 sets of 15 minutes (breathing against 100% of the training load) with 1-min interval between them. Heart rate and BP will be monitored in all training sessions. The RMS, iRME, respiratory constant load tests and CPET will be performed before and after the training, and in the 3rd and 7th week (for training load adjustment). The pulmonary function testing and the cardiovascular autonomic tests will be performed only before and after training. The data will be analyzed by specific statistical tests (parametric and nonparametric) according to the data distribution and their respective variances. Significance will be set at p<0.05. Expected results: It is expected that the training performed by PTHCG, when compared to training performed by 60G and PG, promotes: greater improvementin workload (Watts) and peak oxygen uptake (VO2peak); increasing in MIP and iRME; decreasing of dyspnoea and peripheral fatigue; delay in activation of muscle metaboreflex in the CPET and iRME; improvement incardiac parasympathetic autonomic modulation and reducing cardiac and peripheral sympathetic modulation. Moreover, it is expected that the results can provide information for a better understanding of the responses obtained by the PThC training in the different evaluated systems. In addition, these results will allow the use of this method by health professionals as a new assessment tool and IMT prescription.

ELIGIBILITY:
Inclusion Criteria:

* Apparently Healthy;
* Practicing cycling for at least 6 months continuous and at least 150 min weekly as active [by the American College of Sports Medicine (2011)].

Exclusion Criteria:

* Participants can not be: smokers, alcoholics, illegal drug users or drugs that may interfere in the search results;
* Diagnosis of cardiorespiratory and metabolic disease;
* Absence of ischemic and conduction ECG alterations at rest or during the clinical exercise test;
* Body mass index (BMI) <30 kg/m²;
* Presence of respiratory muscle weakness [maximal inspiratory pressure (MIP <60% predicted);
* Alterations in the pulmonary function test (PFT) or other test;
* Have performed of inspiratory muscle training in the last six months.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Performance in exercise evaluated by measurement the maximal or peak comsumption the oxygen (VO2max or peak) | Three years
  The performance will be evaluated by measurement the maximal or peak comsumption the oxygen (VO2max or peak), determinated by the cardiopulmonary exercise testing.
Performance in exercise evaluated by measurement the work load (W) | Three years
  The performance will be evaluated by measurement the work load (W), determinated by the cardiopulmonary exercise testing.
  The evaluation will realize before, fifth and ninth weeks and after the training.

SECONDARY OUTCOMES:
Cardiovascular responses to inspiratory muscle training | Three years
  The cardiovascular responses [systolic arterial pressure (PAS), dyastolic arterial pressure (PAD), using Finometer PRO; and heart rate, using BioAmp FE132] will be evaluated during the cardiopulmonary exercise testing and progressive inspiratory threshold-loading test, .
  The evaluation will realize before, fifth and ninth weeks and after the training.
Respiratory responses to inspiratory muscle training | Three years
  The ventilatory parameters [carbon dioxide production (VCO₂), respiratory exchange rate (RER), lung ventilation (VE), oxygen uptake efficiency slope (OUES), minute ventilation-carbon dioxide production slope (VE/VCO₂slope)] will monitored and registered breath-by-breath using a ventilatory-metabolic system ULTIMA/Breeze Suite 7.2., during cardiopulmonary exercise test and progressive inspiratory threshold-loading test.
  The evaluation will realize before, fifth and ninth weeks and after the training.
Metabolic responses to inspiratory muscle training | Three years
  The oxyhemoglobin, deoxyhemoglobin and total hemoglobin responses will be measured by near-infrared spectroscopy (NIRS) (Oxymon MKIII), during cardiopulmonary exercise test and progressive inspiratory threshold-loading test.
  The evaluation will realize before, fifth and ninth weeks and after the training.
Autonomic responses to inspiratory muscle training | Three years
  The cardiovascular autonomic tests, heart rate variability (HRV) and blood pressure variability (BPV), at rest and after active postural change will realize before and after the training.
  The ECG (BioAmp FE132), blood pressure (BP), using Finometer Pro (Finapress Medical Systems) and respiration (Marazza) signals will be acquired. The signals will be coupled by data acquisition and analysis device (Power Lab 8/35) and sampled at 1000 Hz.
Metaboreflex activation to inspiratory muscle training | Three years
  To evaluate if the IMT, using PThC, changes the intensity of the metaboreflex activation, evaluated during the cardiopulmonary exercise testing and the progressive inspiratory threshold-loading test.
  The evaluation will realize before, fifth and ninth weeks and after the training.

CONTACTS AND LOCATIONS:
Overall Officials: Aparecida M Catai, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of Sao Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] HajGhanbari B, Yamabayashi C, Buna TR, Coelho JD, Freedman KD, Morton TA, Palmer SA, Toy MA, Walsh C, Sheel AW, Reid WD. Effects of respiratory muscle training on performance in athletes: a systematic review with meta-analyses. J Strength Cond Res. 2013 Jun;27(6):1643-63. doi: 10.1519/JSC.0b013e318269f73f. PMID 22836606
- [Background] Hautmann H, Hefele S, Schotten K, Huber RM. Maximal inspiratory mouth pressures (PIMAX) in healthy subjects--what is the lower limit of normal? Respir Med. 2000 Jul;94(7):689-93. doi: 10.1053/rmed.2000.0802. PMID 10926341
- [Derived] Rehder-Santos P, Minatel V, Milan-Mattos JC, Signini EF, de Abreu RM, Dato CC, Catai AM. Critical inspiratory pressure - a new methodology for evaluating and training the inspiratory musculature for recreational cyclists: study protocol for a randomized controlled trial. Trials. 2019 May 7;20(1):258. doi: 10.1186/s13063-019-3353-0. PMID 31064379